CLINICAL TRIAL: NCT01108861
Title: The GORE VIABAHN® Endoprosthesis With PROPATEN Bioactive Surface Versus Plain Old Balloon Angioplasty (POBA) for the Treatment of Superficial Femoral Artery (SFA) In-Stent Restenosis
Brief Title: GORE VIABAHN® Versus Plain Old Balloon Angioplasty (POBA) for Superficial Femoral Artery (SFA) In-Stent Restenosis
Acronym: RELINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMRP-100107
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral Vascular Disease; In-stent restenosis; Endoprosthesis; Plain old balloon angioplasty
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoprosthesis (Experimental): GORE VIABAHN® Endoprosthesis
  Interventions: Device: GORE VIABAHN® Endoprosthesis
- Plain old balloon angioplasty (Active Comparator): Plain old balloon angioplasty
  Interventions: Device: Plain old balloon angioplasty

INTERVENTIONS:
Device: GORE VIABAHN® Endoprosthesis — GORE VIABAHN® Endoprosthesis
  Arms: Endoprosthesis
Device: Plain old balloon angioplasty — Plain old balloon angioplasty
  Arms: Plain old balloon angioplasty

SUMMARY:
This is a prospective, randomized, multi-center study recruiting patients with an in-stent restenosis in the superficial femoral artery. The safety and efficacity of the Viabahn endoprosthesis (W.L. Gore & Associates), a heparin-bonded endoprosthesis, is compared with plain old balloon angioplasty (POBA). In 4 Belgian and 2 German centers a total of 80 Patients will be recruited. Primary endpoint is primary patency at 12 months, defined as no evidence of restenosis or occlusion within the originally treated lesion based on color-flow duplex ultrasound (CFDU) measuring a peak systolic velocity ratio ≤2.5, and without target lesion revascularization (TLR) within 12 months.

In comparison to POBA, it is expected that the use of the Viabahn endoprosthesis (W.L. Gore & Associates) will result in greater 12 month primary patency of treated superficial femoral artery in-stent restenotic lesions.

ELIGIBILITY:
General Inclusion Criteria:

* Patient presenting with lifestyle-limiting claudication, rest pain or minor tissue loss (Rutherford classification from 2 to 5)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 24 months
* Noninvasive lower extremity arterial studies (resting or exercise) demonstrate ankle-brachial index ≤0.8
* Patient is eligible for treatment with the Viabahn® Endoprosthesis (W.L. Gore)
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure

Angiographic Inclusion Criteria

* Restenotic or reoccluded lesion located in a stent which was previously implanted (>30 days) in the superficial femoral artery, suitable for endovascular therapy
* Total target lesion length between 4 and 27 cm (comprising in-stent restenosis and adjacent stenotic disease)
* Minimum of 1.0cm of healthy vessel (non-stenotic) both proximal and distal to the treatment area
* Popliteal artery is patent at the intercondylar fossa of the femur to P3
* Target vessel diameter visually estimated to be >4mm and <7.6 mm at the proximal and distal treatment segments within the SFA
* Guidewire and delivery system successfully traversed lesion
* There is angiographic evidence of at least one-vessel-runoff to the foot, that does not require intervention (<50% stenotic)

Exclusion criteria :

* Untreated flow-limiting aortoiliac stenotic disease
* Presence of a chronic total occlusion, i.e. a complete occlusion of the failed bare stent that cannot be re-opened with thrombolysis or does not allow easy passage of the guidewire by the physician
* Any previous surgery in the target vessel
* Severe ipsilateral common/deep femoral disease requiring surgical reintervention
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Femoral or popliteal aneurysm located at the target vessel
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* No patent tibial arteries (>50% stenosis)
* Prior ipsilateral femoral artery bypass
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol or 2-year life expectancy
* Serum creatinine >2.5mg/dL within 45 days prior to study procedure unless the subject is currently on dialysis
* Major distal amputation (above the transmetatarsal) in the study or non-study limb
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergies to stent or stent graft components (nickel-titanium or ePTFE)
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial, unless approved by W.L. Gore & Associates in advance of study enrolment
* Angiographic evidence of intra-arterial thrombus or atheroembolism from inflow treatment
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Target lesion access not performed by transfemoral approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months, defined as no evidence of restenosis or occlusion within the originally treated lesion based on color-flow duplex ultrasound (CFDU) and without target lesion revascularization (TLR) within 12 months. | 1 year
Proportion of subjects who experience serious device-related adverse events within 30 days post-procedure | 30 days

SECONDARY OUTCOMES:
Technical success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%. | during procedure
Hemodynamic primary patency rate at 1, 6, 12, 24-month follow-up. | 1, 6, 12, 24-month follow-up
  Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (systolic velocity ratio no greater than 2.5) and without prior TLR are defined as being primary patent at the given follow-up.
Angiographic primary patency at 12 months | 1 year
  Angiographic primary patency at 12 months, defined as no evidence of restenosis or occlusion within the originally treated lesion based on no Quantitative Angiographic evidence of stenosis > 50%
Primary assisted patency rate at 1, 6, 12, 24-month follow-up. | 1, 6, 12, 24-month follow-up
  Primary assisted patency rate at 1, 6, 12, 24-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention completed prior to complete vessel closure.
Secondary patency rate at 1, 6, 12, 24-month follow-up | 1, 6, 12, 24-month follow-up
  Secondary patency rate at 1, 6, 12, 24-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention after occlusion of the target lesion.
Target lesion revascularization (TLR) | entire follow-up
  Target lesion revascularization (TLR) is defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the device/PTA edge
Clinical success at follow-up | at 1 day and 1, 6, 12, 24-month follow-up
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1 day and 1, 6, 12, 24-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Serious adverse events | during entire follow-up
  Serious adverse events as defined as any clinical event that is fatal, life-threatening, results in persistent or significant disability/incapacity, requires in-patient hospitalization or unduly prolonged hospitalization, necessitates an intervention to prevent a permanent impairment of a body function or permanent damage to a body structure, is a congenital abnormality/birth defect, a fetal distress or fetal death, results in malignancy
Stent fracture rate at 12 months | 1 year
  Stent fracture rate at 12 months, determined by using the following classifications on X-ray:
  1. Class 0 : no strut factures
  2. Class I : single tine fracture
  3. Class II : multiple tine factures
  4. Class III : Stent fracture(s) with preserved alignment of the components
  5. Class IV : Stent fracture(s) with mal-alignment of the components
  6. Class V : Stent fracture(s) in a trans-axial spiral configuration

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint Blasius
Locations (6):
- Belgium (4):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - Universitair ziekenhuis antwerpen, Edegem
  - Zuid Oost Limburg, Genk
- Germany (2):
  - Herz-zentrum Bad Krozingen, Bad Krozingen
  - Herzzentrum, Leipzig

REFERENCES:
- [Derived] Bosiers M, Deloose K, Callaert J, Verbist J, Hendriks J, Lauwers P, Schroe H, Lansink W, Scheinert D, Schmidt A, Zeller T, Beschorner U, Noory E, Torsello G, Austermann M, Peeters P. Superiority of stent-grafts for in-stent restenosis in the superficial femoral artery: twelve-month results from a multicenter randomized trial. J Endovasc Ther. 2015 Feb;22(1):1-10. doi: 10.1177/1526602814564385. PMID 25775672